CLINICAL TRIAL: NCT00357006
Title: Multisite Double-Blind Randomized Controlled Study of Estradiol Plus Antipsychotic Versus Placebo Plus Antipsychotic in the Treatment of Psychotic Symptoms in Women With Schizophrenia
Brief Title: A Definitive Estrogen Patch Study (ADEPT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Alfred (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Jayashri Kulkarni, Professor, Director, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202/04; 05T-742
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder(Not in Manic Phase)
Keywords: Schizophrenia; Estrogen; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): 100 mcg Estradiol
  Interventions: Drug: Estradiol
- 2 (Active Comparator): 200 mcg Estradiol
  Interventions: Drug: Estradiol
- 3 (Placebo Comparator): adjunctive transdermal placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Estradiol — 100 mcg adjunctive transdermal estradiol
  Arms: 1
Drug: Estradiol — 200 mcg adjunctive transdermal estradiol
  Arms: 2
Other: placebo — adjunctive transdermal placebo
  Arms: 3

SUMMARY:
OBJECTIVE:

To test the use of adjunctive estrogen in a 8 week, three-arm, double-blind, placebo-controlled study in the treatment of psychotic symptoms in women with schizophrenia.

HYPOTHESIS:

That women receiving adjunctive estrogen will demonstrate significantly greater improvements in the symptoms of schizophrenia than women receiving adjunctive placebo.

STUDY POPULATION:

180 women will be recruited over a three-year period across three sites. Participant will be of potential child-bearing age (Pre-menopausal and Post-menarche) with a current diagnosis of Schizophrenia, Schizophreniform Disorder, or Schizoaffective Disorder (not in manic phase)according to the Mini International Neuropsychiatric Interview (MINI).

STUDY MEDICATION:

Estradiol. One third of the participants (n=60) will be randomised to receive adjunctive 100mcg Estradiol; one third of the participants (n=60) will be randomised to receive adjunctive 200mcg Estradiol n=60; and, one third of the participants (n=60) will be randomised to receive adjunctive placebo n=60). All patches will be covered with identical adhesive contact to ensure the "blind" is maintained.

STUDY EVALUATIONS:

Data will be collected over a two-month period for each participant. Visits will be performed at baseline, and then at weekly or fortnightly intervals. A total of six visits will be completed for each participant. The following evaluations will be performed:

i) Inclusion/exclusion checklist. (Baseline visit only)

ii) Informed consent. (Baseline visit only)

iii)psychiatric evaluation to determine diagnosis. (Baseline visit only)

iv) General clinical evaluation including medical history, current conditions and a non-invasive physical examination, body weight, vital signs. (Baseline and endpoint visits)

v) Medication history. (Baseline and evaluation visits)

vi) Demographics. (Baseline visits only)

vii) The primary outcome measures will be the Positive and Negative Syndrome Scale (PANSS), which will be taken at weeks 1, 2, 4 and 8 of the trial. Cognitive testing will take place at baseline and 8 weeks. Side effects will be assessed at weeks 1, 2, 4, 6, and 8 to measure changes in subject's reported side effects during the trial.

viii) Laboratory tests including; Serum levels of mood stabiliser, LH, FSH, Estrogen, Progesterone, Prolactin, DHEA,Testosterone and(Baseline and evaluation visits).

DETAILED DESCRIPTION:
This research protocol outlines a multi-site clinical trial of adjunctive estradiol in women with Schizophrenia. We propose to recruit 180 women into this study from 3 Australian sites - The Alfred Hospital, Barwon Health, and Dandenong Hospital.

1.1 Literature Review

Schizophrenia is a severe mental disorder that affects up to 2% of the adult population. Patients present with a variety of symptoms including hallucinations, delusions and bizarre behaviour while some develop additional "negative" symptoms such as amotivational states and poverty of thought.

Schizophrenia is generally thought to be an organic brain disorder with psychosocial determinants for course and outcome. The illness appears to be heterogenous with groups of patients presenting with distinct and differing patterns of psychopathology and illness course. Part of this heterogeneity includes distinct male and female subtypes of schizophrenia.

In recent times, gender differences in schizophrenia have received some attention, in particular from an epidemiological and psychopathological perspective. Hormonal studies have been utilised to investigate underlying neuroendocrine disturbances in schizophrenia, but information from these studies has not been used in the development of new gender specific treatment strategies. Overall the treatment of schizophrenia has remained gender-blind. The main gender differences observed in schizophrenia that have international consensus include the later age of onset in women; better response to antipsychotics in women; and more treatment resistant negative symptoms in men. Women have also demonstrated vulnerability to psychotic episodes during menopause, the post-partum period and at low estrogen phases of the menstrual cycle.

From these clinical observations, Seeman and Lang (1990) hypothesised that estrogen may provide "protection" against early onset of severe schizophrenia in women, thereby accounting for increased vulnerability during both lifetime and monthly low estrogen phases. Seeman and Lang (1990) further hypothesised that estrogen may provide protection against early onset of severe treatment resistant schizophrenia through an anti-dopaminergic effect by modulating the sensitivity of the dopamine receptor thereby potentiating the effect of antipsychotics.

Evidence for estrogen having a modulating effect on dopaminergic systems comes from studies in rats in which estrogens can enhance antipsychotic-induced cataplexy (Behrens et al. 1992; Fields et al 1982) and reduce amphetamine and apomorphine-induced behaviour such as stereotypies (Ferretti et al., 1992; Clopton et al., 1986). In humans, the presence of estrogen receptors in the limbic system indicates that estrogens may have a neuromodulatory function (Foreman, et al., 1980; Koller, et al., 1980; Gordon et al., 1980). Estrogens have been shown to reduce the dopamine concentration in the striatum (Dupond et al., 1981; Bedard et al., 1984) and modulate the sensitivity as well as the number of dopamine receptors (Di Paolo, et al., 1981; McDermott, et al., 1994). There are clinical case reports of women whose schizophrenic symptomatology is exacerbated at low estrogen phases of the menstrual cycle (Endo et al., 1978). Similarly there are clinical case reports of women with chronic schizophrenia improving during pregnancy - when estrogen levels are extremely high (Seeman, 1986). After delivery, when estrogen levels drop, increased vulnerability to psychosis is observed (Seeman, 1996). A recent study investigating the relationship between schizophrenia psychopathology and low estrogen phases of the menstrual cycle revealed that symptoms improved when natural estradiol levels increased (Riecher-Rossler et al., 1994). This study also showed that all 32 patients studied had markedly reduced serum estradiol levels compared with the normal population and that fluctuations throughout the cycle were dampened.

1.2 Justification for Project

The findings from both basic and clinical research reviewed in section 1.1 above warrant further investigation of the hypothesis that estrogen has a protective effect in women, not only over the female life cycle, but also over the menstrual cycle. Case reports have appeared in the literature in which clinicians detail improvement in one or two female patients following administration of synthetic combined estrogen and progesterone. A study conducted by Klaiber and colleagues' (1979) reported that large doses of estrogen assisted in the treatment of depression in women. We have been conducting clinical trials in patients with schizophrenia using estrogen as a treatment for many years, and have an international reputation for work in this area. Initially, we conducted an open clinical trial with acutely ill schizophrenic women (Kulkarni et al., 1996) and added 0.02mg of oral estradiol to the antipsychotic drug treatment of 11 women. Their response was compared to seven women who received antipsychotic drugs alone. The estrogen adjunct group showed dramatic earlier improvement, with significant reduction in positive psychotic symptoms by day 3 of treatment. This suggests that estradiol may act as a catalyst for treatment and could prove to be an important adjunctive treatment in the therapy of schizophrenia. Subsequent to this early pilot study, we conducted a double blind placebo controlled 3-arm study of 100mcg, 50mcg estradiol and placebo transdermal adjunctive patches. Published in Schizophrenia Research (Kulkarni et al., 2003), our results showed that the 100mcg estrogen adjunct afforded the best outcomes. We then conducted a "proof of concept" study to examine the effect of adding 100mcg transdermal estrogen versus transdermal placebo to antipsychotic drug treatment in 90 women with schizophrenia. For the results of this 'proof of concept' study please refer to Appendix G.

1.3 Review of Estradiol and its Uses

Estrogen is one of a group of hormonal steroid compounds that promote the development of female secondary sex characteristics. Human estrogen is produced by the ovaries, adrenal cortices, testes, and feto-placental unit. Along with progesterone, estrogen plays a major role in the regulation of the menstrual cycle and is regulated by levels of Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH) released from the anterior pituitary gland in the brain. These two gonadotropin hormones are in turn regulated by the actions of the hypothalamus. Pharmaceutical preparations of estrogen are used in oral contraceptives, to palliate post-menopausal breast cancer and prostatic cancer, to inhibit lactation, and to treat threatened abortion, osteoporosis and ovarian disease. Estrogen is also given to relieve the discomforts of menopause. Types of estrogen are conjugated estrogen, esterified estrogen, estradiol, estriol and estrone (Mosby, 1986). Delivery of estrogen by transdermal patches provides more natural and physiologically equivalent replacement of estradiol levels.

2. RESEARCH OBJECTIVES

To conduct a three-arm, double-blind, randomized, placebo-controlled, trial across three sites, to investigate the 'estrogen-protection' hypothesis in women with schizophrenia. The study aims to:

1. replicate previous research, thereby providing 'proof of concept' for the potential use of estradiol as a treatment in women with schizophrenia;
2. investigate the effect of an increased dose of estradiol (200mcg transdermal);
3. investigate the duration of the "antipsychotic effect" of estradiol

   The aims will be met by comparing changes in psychopathology and cognition over an 8-week period between three groups of participants: (1) a group of participants receiving standard antipsychotic treatment and a placebo; (2) a matched group receiving standard antipsychotic treatment plus 100mcg estradiol patches; and (3) a matched group receiving standard antipsychotic treatment plus 200mcg estradiol patches.

   3. ETHICS REVIEW AND INFORMED CONSENT

   3.1 Ethics Review

   The protocol for this study was approved by the Alfred Research & Ethics Committee on 6th January 2005, at the Barwon site on 01/03/2006, and at the Dandenong site on 12/05/2006.

   3.2 Issues Related to the Use of Estradiol Skin Patches

   The study involves the addition of 100mcg/200mcg estradiol to standard antipsychotic treatment for 8 weeks. This dose of estradiol is commonly used in hormone replacement therapy for postmenopausal women, without side effects. The length of the trial is 2 menstrual cycles, which is a short period of estrogen use. Most side effects commonly associated with estrogen use are related to long term administration and are thus not applicable in this study. Basic medical precautions will be taken prior to the commencement of estrogen therapy (ie. physical examination, routine investigations and pregnancy testing). In our large study of 90 women 100mcg transdermal estradiol was used and the treatment was well tolerated. Subjects will be counselled with regard to the lack of contraceptive effect of using estradiol patches.

   3.3 Use of a Placebo

   All subjects will be informed that there is a two-in-three chance that they will receive estradiol patches and a one-in-three chance they will receive placebo patches. As well as the study medication, all subjects will receive standard antipsychotic medication and thus will not be disadvantaged in any way by placement in the "placebo" group. Subjects who are entered into the trial will be on a relatively stable treatment regime having had no change of medication in the prior 30 days and there will be no future change in medication anticipated. By controlling this variable, we are able to create a 'true placebo' group as there should be no modification of antipsychotic medication over the trial period that could potentially affect the psychopathology results. Both subjects and researchers will be unaware of which group a subject is in. However, if the need arises researchers will be able to break the code to reveal the group to which the subject belongs. Subjects allocated to the placebo group will be offered open-label adjunctive treatment with 200mcg estradiol for two months proceeding the trial, thereby ensuring all participants receive the potential benefits of adjunctive estradiol.

   3.4 Standard Antipsychotic Treatment

   As the proposed study is an adjunctive trial, all participants will continue to receive standard antipsychotic treatment whilst in the trial. Antipsychotic medication will be measured in "risperidone equivalents", which involves converting the dose of their current antipsychotic treatment to its equivalent dose of risperidone. To be included in the trial participants must meet the following criteria: 2-10mg daily "risperidone equivalents" for at least 4 weeks with residual symptoms as defined by a PANSS positive score greater than 15 and/or a PANSS negative score greater than 15.

   3.5 Informed Consent

   Only participants who are able to give informed consent, i.e. able to demonstrate an understanding of the objectives of the study and the implications of their role in it, will be recruited into the study. Involuntary patients who are able to give informed consent will be able to participate and where possible a guardian or relative will be contacted and notified of the patients' involvement. Participants will be advised that their participation is voluntary and that they are free to withdraw from the study at any stage.

   3.6 Confidentiality

   Participants' identity will remain anonymous at all times. Once a participant agrees to participate in the study, she will be assigned a code number to ensure anonymity. Information about the subject will be restricted to the researchers directly involved, unless there are clear management issues, in which case the information will be shared with the treatment team. Participants' files will be stored in locked filing cabinets with access only available to researchers on the project. All test results will be shared with the participant and their family / guardian.

   4. METHOD

   4.1 Participants

   A target number of 180 participants (60 from The Alfred, 60 from Barwon and 60 from Dandenong) will be recruited over a three-year period with equal numbers being allocated to each group (100mcg Estradiol n=60; 200mcg Estradiol n=60; Placebo n=60). Participants will be recruited from both inpatient and outpatient settings and participants may be recruited from other centres providing that approval has been gained from the appropriate controlling bodies. The total number of subjects will allow results to be analysed by subgroups based on factors such as menstrual cycle phase.

   4.2 Materials
   * demographic information
   * diagnosis according to the Mini International Neuropsychiatric Interview (MINI) - modules L (psychotic disorders) and D (mania/hypomania )
   * inclusion/exclusion criteria check
   * medical history & non-invasive general physical examination
   * Laboratory tests to determine pregnancy status, menstrual cycle phase and neuroendocrine status
   * Breast scan (mammogram; at Alfred and Dandenong sites) or breast screens (ultrasounds; at Barwon site) to check for breast abnormalities in participants to be conducted when informed consent is provided
   * hormone measurements of estrogen, progesterone, prolactin, testosterone, LH, FSH and DHEA
   * A menstrual cycle questionnaire (MCQ) to gain a menstrual history
   * Assessment of psychopathology (PANSS & MADRS) and cognitive function (RBANS)

   Hormone assays will be repeated at weeks 4 and 8. A menstrual calendar will be used to record the onset and cessation of menses during the trial. The primary outcome measures will be the Positive and Negative Syndrome Scale (PANSS), which will be taken at weeks 1, 2, 4 and 8 of the trial. Cognitive testing will take place at baseline and 8 weeks. Side effects will be assessed at weeks 1, 2, 4, 6, and 8 to measure changes in subject's reported side effects during the trial.

   4.3 Procedures

   Participants will be screened as soon after identification as possible to assess eligibility for entry into the study. The diagnostic instrument to be used will be the Mini International Neuropsychiatric Interview (MINI). The details of the project and requirements of participation will be explained to eligible participants and a Plain Language Statement provided. If a potential participant is identified to be a current client of The Alfred Psychiatric Service, Southern Health (Dandenong site) or Barwon Health (Barwon site), the researcher will contact a member of the individual's treating team to discuss the suitability of approaching the client and to gain an indication of the person's ability to give informed consent. A member of the treating team will then approach the potential participant and ask if they are willing to talk to the researcher about the study. This discussion will involve providing a detailed verbal explanation of the study and the written Participant Information and Consent Form (PI&CF) as approved by the applicable Human Research Ethics Committee. The potential participant will be asked to read through the PI&CF or have it read to them by the researcher. The potential participant will be encouraged to discuss the PI&CF and the possibility of participating in this study with a significant other or support person.

   Once the potential participant has read the PI&CF the researcher will have another discussion with this person, preferably in the presence of a witness. The researcher will ask the potential participant to provide a verbal explanation about what they think the study is about and what is involved in their participation. The researcher may draw attention to particular parts of the PI&CF to ensure that the potential participant is fully aware of all aspects involved. The potential participant will be asked if he/she has any questions about the study, which will be answered by the researcher. At this point, if the researcher believes that the potential participant understands the information provided to them about the study, and has had the opportunity to ask questions and have them answered, then the consent form can be signed. The consent form will be signed and dated by the project participant, by the researcher who explained the project to the participant, and by a witness.

   Participants who provide informed, written consent will undergo a full psychiatric and medical history and will receive a non-invasive physical examination as well as a breast scan or screen (dependant on site specific regulatory advice). Baseline hormone levels will be measured via a blood test, and a menstrual cycle questionnaire will be administered to determine menstrual status. Baseline psychopathology rating scales (PANSS) will then be administered. After a participant has been deemed eligible to enter the trial and baseline measurements have been performed, the participant may be randomised to one of three groups for the duration of the eight-week double blind phase. The three groups are: (1) 100mcg estradiol patches, (2) 200mcg estradiol patches, and (3) placebo patches.

   Upon entry into the double-blind phase, each participant will be allocated an identification number and will be randomly assigned to a treatment regimen as generated by The Alfred Clinical Trials Pharmacy, who will be aware of which treatment group the participant is allocated to but will not be directly involved in the trial. The Clinical Trials Pharmacy coordinator will not disclose the randomisation codes to any of the investigators or data collectors involved with the project.

   Day one of the trial will be the first day that the participant receives the study medication. Study medication is dispensed via the pharmacy department at each site. Baseline measurements must be taken the day before the first day of the trial, and thus baseline is considered to be Day 0. Evaluation of adverse events and medication compliance will be performed at regular intervals for the duration of the trial. Psychopathology rating scales will be completed at baseline and weeks 1, 2, 4 and 8. Hormone assays will be completed at baseline and weeks 4 and 8. Cognitive assessment will be completed at baseline and at week 8. The week 8 visit must fall on the last day of the trial medication.

   4.4 Clinical Follow-up

   For ethical reasons, upon completion of the active phase of the trial each participant will be "unblinded" and made aware of which treatment they had received. Participants who were receiving placebo will be offered an "open label" trial of the 200mg estradiol patches. This is so that no one is disadvantaged by their participation in the trial and are all able to take the active medication if they so wish. Participants who opt to have an "open label" trial of the estradiol patches will be monitored for side effects for a further 8 weeks whilst they are using the patches. This data will not be included in the research trial database.

   All participants will be followed up for 3 months following the completion of the active phase of the trial (including the open-label treatment). This follow-up will consist of monthly telephone contact to check participant's progress as well as determine the duration of the "antipsychotic effect" of estrogen.

   5. STUDY MANAGEMENT

   5.1 Data Management

   Source data from each site will be transferred to The Alfred site for data entry and analysis. A copy of the source data for each site will be archived at each site according to local ethics committee guidelines. A Contract Research Organisation (CRO) will monitor each of the sites to ensure high quality data and adherence to study recruitment and retention targets. Inter-rater reliability training will be performed annually for all staff at each site or when new staff commence.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of potential child-bearing age (Pre-menopausal and Post-menarche)
* Female participants who meet the MINI (Mini International Neuropsychiatric Interview for DSM-IV) diagnostic criteria for current psychotic disorder or have a current DSM-IV diagnosis of Schizophrenia, Schizophreniform Disorder, or Schizoaffective Disorder (not in manic phase).
* Female participants with a PANSS positive score greater than 15 and/or a PANSS negative score greater than 15.
* Female participants who are able to give informed consent
* Female participants receiving 2-20mg daily Risperidone equivalents for at least 4 weeks.

Exclusion Criteria:

* Female participants who are pregnant or lactating.
* Female participants with known severe abnormalities in the hypothalamo-pituitary gonadal axis, thyroid dysfunction, central nervous system tumours, history of thromboembolic disorders, severe renal failure, severe hepatic failure, cardiac disease, epilepsy or other serious medical conditions which would contraindicate estrogen use.
* Female participants already taking oral estrogen preparations containing greater then 30mcg estradiol.
* Post-menopausal or pre-menarche female participants.
* Female participants whose psychotic illness meets DSM-IV criteria for substance-induced psychotic disorder.
* Female participants who have a current diagnosis of Schizoaffective Disorder and are in a manic phase.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2006-07; Primary Completion 2011-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Kulkarni, MBBS, MPM, FRANZCP, PhD, Principal Investigator — Bayside Health / Monash University
Locations (1):
- Bayside Health - The Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Thomas N, Gurvich C, Hudaib AR, Gavrilidis E, de Castella RA, Thomas EH, Kulkarni J. Serum estradiol as a blood-based biomarker predicting hormonal treatment outcomes in women with schizophrenia. Psychoneuroendocrinology. 2021 Apr;126:105165. doi: 10.1016/j.psyneuen.2021.105165. Epub 2021 Feb 10. PMID 33609856
- See also: Monash Alfred Psychiatry Research Centre — http://www.maprc.org.au/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2006 and 2011, a total of 1858 women were assessed for eligibility, of which 204 were screened from inpatient and outpatient settings across three Australian sites (Alfred, a tertiary referral centre; Barwon, a rural centre; and Dandenong, an outer metropolitan centre) over a 5-year period and completed a 56-day trial.
Groups:
- Adjunctive 200 mcg Transdermal Estradiol: Participants received daily 200mcg transdermal estradiol for 56 days.
- Adjunctive 100 mcg Transdermal Estradiol: Participants received daily 100mcg transdermal estradiol for 56 days.
- Placebo: Participants received daily transdermal placebo for 56 days.
Period: Overall Study
Arm/Group | Adjunctive 200 mcg Transdermal Estradiol | Adjunctive 100 mcg Transdermal Estradiol | Placebo
Started | 62 | 56 | 62
Completed | 60 | 51 | 59
Not Completed | 2 | 5 | 3
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adjunctive 200 mcg Transdermal Estradiol | Adjunctive 100 mcg Transdermal Estradiol | Placebo | Total
Number analyzed (Participants) | 62 | 56 | 62 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 62 | 56 | 62 | 180
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.29 (8.14) | 34.77 (7.28) | 35.44 (8.46) | 35.18 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 56 | 62 | 180
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 62 | 56 | 62 | 180

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: The Positive and Negative Syndrome Scale (PANSS) is a well validated, standardized method of evaluating and monitoring psychotic symptoms. The PANSS assesses: positive (hallucinations, delusions, thought disorder), negative (blunted affect, abstract thinking and general symptomatology. The positive and negative subscale each consist of 7 items rated from 1(absent) - 7(extreme) with a minimum score = 7, maximum score = 49. The general subscale consists of 16 items with a minimum score = 16, maximum score = 112. A Total PANSS score (positive+ negative + general scores) has a minimum of 30 and maximum of 210. Higher scores represent more severity in symptoms.
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Adjunctive 200 mcg Transdermal Estradiol: Participants received daily 200 mcg transdermal estradiol for 56 days.
- Adjunctive 100 mcg Transdermal Estradiol: Participants received daily 100 mcg transdermal estradiol for 56 days.
Arm/Group | Adjunctive 200 mcg Transdermal Estradiol | Adjunctive 100 mcg Transdermal Estradiol | Placebo
Number analyzed (Participants) | 62 | 56 | 62
units on a scale
  Baseline | 18.24 (5.66) | 19.18 (5.54) | 18.18 (5.70)
  Endpoint (day 56) | 14.11 (4.94) | 16.36 (5.57) | 16.36 (5.39)

2. Secondary Outcome: Cognitive Performance (RBANS Scores)
Time Frame: baseline and week 8
Reporting Status: Not Posted

3. Secondary Outcome: Scores on MADRS at Trial Completion
Time Frame: Baseline and week 8
Reporting Status: Not Posted

4. Secondary Outcome: Scores on Adverse Symptom Checklist at Trial Completion
Time Frame: Baseline and weeks 1, 2, 4, 6, 8
Reporting Status: Not Posted

5. Secondary Outcome: Change in Hormone Levels Over Trial Duration
Time Frame: Baseline and weeks 1, 4 and 8.
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Side effects were monitored using an Adverse Symptom Checklist that assesses 18 medication-related adverse effects (nausea, headaches, increased saliva, sexual dysfunction). The Simpson Angus Rating Scale for Extrapyramidal Side Effects, and the Abnormal Involuntary Movement Scale were assessed at each time point (days 0, 7, 14, 28 and 56).
Groups:
- Adjunctive 200 mcg Transdermal Estradiol: Participants received daily 200mcg transdermal estradiol for 8 weeks (56 days).
- Adjunctive 100 mcg Transdermal Estradiol: Participants received daily 100mcg transdermal estradiol for 8 weeks (56 days).
- Placebo: Participants received daily transdermal placebo for 8 weeks (56 days).
Arm/Group | Adjunctive 200 mcg Transdermal Estradiol | Adjunctive 100 mcg Transdermal Estradiol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/56 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/56 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No